CLINICAL TRIAL: NCT00864890
Title: Single Dose Crossover Comparative Bioavailability Study of Citalopram 40 mg Tablets in Healthy Male Volunteers/Fed State
Brief Title: A Relative Bioavailability Study of Citalopram 40 mg Tablets Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Responsible Party: Meena Venugopal, Director, Clinical R&D, Actavis Inc
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: CTA-P2-260
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2010-08-17 (Estimated); Status verified 2010-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Citalopram; Healthy subjects
MeSH Terms: interventions — Citalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): Citalopram HBr 40 mg tablets, single dose
  Interventions: Drug: Citalopram HBr 40 mg tablets, single dose
- B (Active Comparator): CelexaTM 40 mg tablets, single dose
  Interventions: Drug: CelexaTM 40 mg tablets, single dose

INTERVENTIONS:
Drug: Citalopram HBr 40 mg tablets, single dose — A: Experimental Subjects received Purepac formulated products under fed conditions
  Other Names: Citalopram
  Arms: A
Drug: CelexaTM 40 mg tablets, single dose — B: Active comparator Subjects received Forest Labs formulated products under fed conditions
  Other Names: Citalopram
  Arms: B

SUMMARY:
The purpose of this study is to evaluate and compare the relative bioavailability, and therefore the bioequivalence of two formulations of Citalopram after a single dose administration under fed conditions.

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Randomized, 2-period, 2-sequence, crossover design.

Official Title: Single Dose Crossover Comparative Bioavailability Study of Citalopram 40 mg Tablets in Healthy Male Volunteers/Fed State

Further study details as provided by Actavis Elizabeth LLC:

Primary Outcome Measures:

Rate and Extend of Absorption

ELIGIBILITY:
Inclusion Criteria:

1. Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by the informed consent form duly signed by the subject.
2. Males aged from 18 to 50 years with a body mass index (BMI) within 19-30; demographic data (sex, age, ethnic group, body weight, height and smoking habits) will be recorded and reported in the final report.
3. Clinical laboratory values within the laboratory's stated normal range; if not within this range, they must be without any clinical significance and must be recorded as such in the CRF.
4. Healthy according to the laboratory results and physical examination
5. Normal cardiovascular function according to ECG.
6. Subjects should be non- or ex-smokers.

Exclusion Criteria:

1. Significant history of hypersensitivity to citalopram or any related products as well as severe hypersensitivity reactions (like angioedema) to any drugs.
2. Presence or history of significant gastrointestinal, liver or kidney disease, or any other conditions known to interfere with the absorption, distribution, metabolism or excretion of drugs or known to potentiate or predispose to undesired effects.
3. Presence or history of significant cardiovascular, pulmonary, hematologic, neurologic, psychiatric, endocrine, immunologic or dermatologic disease.
4. Use of MAO inhibitors within 14 days of day 1 of the study
5. Maintenance therapy with any drug, or significant history of drug dependency, alcohol abuse (> 3 units of alcohol per day, intake of excessive alcohol, acute or chronic), or serious Psychological disease.
6. Any clinically significant illness in the previous 28 days before day 1 of this study.
7. Use of enzyme-modifying drugs in the previous 28 days before day 1 of this study (all barbiturates, corticosteroids, phenylhydantoins, etc.).
8. Participation in another clinical trial in the previous 28 days before day 1 of this study.
9. Donation of 500 mL or more of blood (Canadian Blood Services, Hema-Quebec, clinical studies, etc.) in the previous 56 days before day 1 of this study.
10. Positive urine screening of drugs of abuse.
11. Positive results to HIV, HBsAg or anti-HCV tests
12. History of fainting upon blood sampling

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2003-06; Primary Completion 2003-07 (Actual); Study Completion 2003-07 (Actual)

PRIMARY OUTCOMES:
Rate and Extend of Absorption | 168 hours

CONTACTS AND LOCATIONS:
Overall Officials: Eric Sicard, M.D., Principal Investigator — Algorithme Pharma Inc
Locations (1):
- Algorithme Pharma Inc., Montreal, Quebec, Canada